CLINICAL TRIAL: NCT01824134
Title: A Phase III Double Blind Study on the Efficacy of Topical Aloe Vera Gel on Irradiated Breast Tissue
Brief Title: Aloe Vera on Irradiated Breast Tissue
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: John D. Archbold Memorial Hospital (Other)
Responsible Party: Principal Investigator, J. Steven Johnson, MD, J. Steven Johnson, MD, John D. Archbold Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 12-09-008
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Irradiated Breast Tissue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Klean & Klear (Active Comparator): aloe vera gel
  Interventions: Other: Klean & Klear The Dandy Day Corp
- The Skin Gel (Active Comparator): aloe vera gel
  Interventions: Other: The Skin Gel Herbal Answers, Inc

INTERVENTIONS:
Other: Klean & Klear The Dandy Day Corp
  Arms: Klean & Klear
Other: The Skin Gel Herbal Answers, Inc
  Arms: The Skin Gel

SUMMARY:
The investigators are testing two over the counter aloe veras on irradiated breast tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Women over 18 years of age who had undergone lumpectomy or partial mastectomy for breast cancer, and who then received postoperative radiation therapy using tangential fields, with or without a boost to the tumor bed. Chemotherapy as part of the treatment regimen was acceptable.
2. No major medical or psychiatric illness that might interfere with patient's completion of study requirements
3. Signed study-specific informed consent form prior to study entry

Exclusion Criteria:

1. Those requiring nodal radiation therapy were excluded.
2. Subjects who have a breast infection at the commencement of radiation treatment
3. Before randomization, subjects who have agreed to participate are asked if they are allergic to any topical preparation. Those allergic to aloe vera were ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
erythema | one year
  since we are testing two over the counter products we wanted to wee if one tested better than the other

SECONDARY OUTCOMES:
itching | one year
  is there a difference in itching

CONTACTS AND LOCATIONS:
Locations (1):
- Lewis Hall Singletary Oncology Center at John D. Archbold Memorial Hospital, Thomasville, Georgia, United States